CLINICAL TRIAL: NCT00367887
Title: A Phase 2, Randomized, Open-Label Study Of The Safety, Antiviral Activity, And Pharmacokinetics Of HCV-796 Administered In Combination With Peginterferon Alfa 2B (Peg-Intron) Plus Ribavirin (Rebetol) Versus Peg-Intron Plus Rebetol In Subjects With Hepatitis C Virus Genotype 1 Infection
Brief Title: A Study Evaluating the Safety and Clinical Activity of HCV-796 in Treatment-Naive and Non-Responder Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Collaborators: ViroPharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3173A1-200; B3381001
Record Dates: First submitted 2006-08-21; First posted 2006-08-23 (Estimated); Last update posted 2013-02-11 (Estimated); Status verified 2013-02

CONDITIONS: Hepatitis C
Keywords: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — peginterferon alfa-2b; Ribavirin; HCV 796

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator)
  Interventions: Drug: Peg-Intron; Drug: REBETOL
- 2 (Active Comparator)
  Interventions: Drug: HCV 796; Drug: Peg-Intron; Drug: REBETOL
- 3 (Active Comparator)
  Interventions: Drug: HCV 796; Drug: Peg-Intron; Drug: REBETOL

INTERVENTIONS:
Drug: Peg-Intron — SC injection, weight based dosing, weekly, 48 weeks
  Arms: 1
Drug: REBETOL — Capsules, weight based dosing, Q12 hrs daily, 48weeks
  Arms: 1
Drug: HCV 796 — Capsules, 500 mg, Q 12 hrs. daily, 48 weeks
  Arms: 2
Drug: Peg-Intron — SC injection, weight based dosing, weekly, 48 weeks
  Arms: 2
Drug: REBETOL — Capsules, weight based dosing, Q12 hrs daily, 48weeks
  Arms: 2
Drug: HCV 796 — Capsules, 500 mg, Q 12 hrs. daily, 48 weeks
  Arms: 3
Drug: Peg-Intron — SC injection, weight based dosing, weekly, 48 weeks
  Arms: 3
Drug: REBETOL — Capsules, weight based dosing, Q12 hrs daily, 48weeks
  Arms: 3

SUMMARY:
This is a phase 2, randomized, open-label study comparing the safety, antiviral activity, and pharmacokinetics of HCV-796 administered in combination with peginterferon alfa 2B (Peg-Intron) plus concomitant Rebetol vs. Peg-Intron plus Rebetol in Hepatitis C Virus (HCV) genotype

1-infected subjects who are either naive to treatment or who have previously failed treatment (non-responders).

ELIGIBILITY:
Inclusion Criteria:

* Infection with HCV genotype 1.
* HCV- infected subjects naive to treatment.
* HCV-infected non-responder subjects.

Exclusion Criteria:

* Women who are pregnant or breastfeeding.
* ALT >/ or = 5X the upper limit of normal.
* AST >/ or = 5X the upper limit of normal.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Actual)
Dates: Start 2006-10; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Hepatitis C Virus (HCV) RNA concentrations in the blood. | 72 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (30):
- United States (29):
  - Pfizer Investigational Site, Anaheim, California
  - Pfizer Investigational Site, La Jolla, California
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, Pasadena, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, San Francisco, California
  - Pfizer Investigational Site, Washington D.C., District of Columbia
  - Pfizer Investigational Site, Gainesville, Florida
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, Louisville, Kentucky
  - Pfizer Investigational Site, Boston, Massachusetts
  - Pfizer Investigational Site, Worcester, Massachusetts
  - Pfizer Investigational Site, Detroit, Michigan
  - Pfizer Investigational Site, Plymouth, Minnesota
  - Pfizer Investigational Site, Saint Paul, Minnesota
  - Pfizer Investigational Site, St Louis, Missouri
  - Pfizer Investigational Site, Albuquerque, New Mexico
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, The Bronx, New York
  - Pfizer Investigational Site, Chapel Hill, North Carolina
  - Pfizer Investigational Site, Durham, North Carolina
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, Cleveland, Ohio
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, Annandale, Virginia
  - Pfizer Investigational Site, Fairfax, Virginia
  - Pfizer Investigational Site, Richmond, Virginia
- Pfizer Investigational Site, Santurce, Puerto Rico

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3173A1-200&StudyName=A%20Study%20Evaluating%20the%20Safety%20and%20Clinical%20Activity%20of%20HCV-796%20in%20Treatment-Naive%20and%20Non-Responder%20Subjects